CLINICAL TRIAL: NCT04028882
Title: Immune Activation as a Cause of Insulin Resistance in Adults Living With HIV-1 on Effective Antiretroviral Therapy
Acronym: MetACTIVIH
Status: Terminated | Type: Observational
Why Stopped: Preliminary analyses regarding the main objective show negative results
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0373
Record Dates: First submitted 2019-06-12; First posted 2019-07-23 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Signal Transduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and peripheral blood mononuclear cells (PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non viremic HIV patients under treatment: Patients with various immune activation profiles
  Interventions: Other: Signaling, metabolomic and transcriptomic analysis

INTERVENTIONS:
Other: Signaling, metabolomic and transcriptomic analysis — Signaling, metabolomic and transcriptomic analysis

SUMMARY:
The aim of this study is to characterize in non-viremic HIV-1 patients under antiretroviral therapy an immune activation profile that the investigators have previously shown to be strongly linked to hyperinsulinemia. This characterization will be carried out via 3 different approaches. First, the investigators will analyze the metabolites present in the plasma of patients presenting with the profile of interest. Second, the investigators will study the transcriptome of the peripheral blood mononuclear cells of these patients. Finally, the investigators will search whether some factors released by these cells are able to induce insulin resistance. In addition the ability of the profile of interest to predict an increase in insulinemia over time will be assessed.

DETAILED DESCRIPTION:
The working hypothesis of this study is that in efficiently treated HIV patients, various profiles of immune activation may be distinguished, each favouring particular comorbidities. Using a panel of 68 soluble and cell surface markers, the investigators have previously measured the level of activation in circulating Cluster of Differentiation 4+ (CD4+) and Cluster of Differentiation 8+ (CD8+), T cells, B cells, monocytes, Natural Killers (NK) cells, neutrophils, and endothelial cells as well as of inflammation and fibrinolysis in 120 virologic responders over 45 years of age. Two independent hierarchical clustering analyses allowed the investigators to identify five patient groups, each with the same activation profile. One of these profiles, Profile#2, was strongly associated with hyperinsulinemia (Psomas et al., 2016).

The main objective of the present study is to better define Profile#2. To this aim, the investigators will analyze by mass spectrometry the metabolites in the plasma of patients with various profiles including the one of interest. Concurrently, the investigators will perform an RiboNucleic Acid Sequencing (RNASeq) analysis on peripheral blood mononuclear cells (PBMC) from the same patients. These metabolomic and transcriptomic data will help to better define the immune activation profiles.

The secondary objective is to test whether the link the investigators have observed between Profile#2 and insulin resistance is causative. To this aim, by following over time patients' insulinemia, the investigators will test whether Profile#2 is predictive of an increase in insulinemia. The investigators will also look for factors released by PBMC of patients with Profile#2 able to induce insulin resistance.

ELIGIBILITY:
Inclusion criteria:

* Subject consulting or hospitalized in the tropical and infectious diseases unit at the University Hospital of Montpellier that have been enrolled in a study during which the immune activation profile was analyzed
* Subject aged at least 18 years
* Subject speaking french fluently
* Subject who is not opposed to participate to the study, after a clear information
* Subject affiliated to a social security system
* Infection by HIV-1 determined by a positive serology or by a measure of the plasma viral load (RNA HIV)
* HIV-1 patients under stable antiretroviral therapy
* HIV load < 50 copies/mL since at least 6 months before enrollment (2 measures)

Exclusion criteria:

* Vulnerable individuals
* Persons protected
* Pregnant women or breastfeeding mothers
* Bad understanding of the nature and goals of the study and/or communication difficulties with the investigator
* Subject enrolled in an other study with an exclusion period still running
* Non infectious pathology that might be the origin of an immune anomaly
* Treatment by an immune modulator molecule or by chemotherapy in the 60 days before enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1-infected adults under efficient antiretroviral therapy
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Metabolomic analysis on plasma and PBMC | 18 months
  The investigators will analyze by mass spectrometry the metabolites present in the plasma of patients presenting with the profile of interest as compared with patients with other immune activation profiles. Metabolites will be extracted from the blood plasma using a salt assisted liquid-liquid extraction. The metabolites will then be allowed to crystallize on the metallic surface. Finally, the plate content will be analyzed by desorption electrospray ionisation mass spectrometry using positive and negative ionization.
Transcriptomic analysis on plasma and PBMC | 18 months
  The investigators will also analyze by RNASeq the messenger RNA (mRNA) produced by the PBMC of patients presenting with the profile of interest and compared them with the mRNA produced by the PBMC of patients with other immune activation profiles.

SECONDARY OUTCOMES:
Follow-up over time of insulinemia in patients with various immune activation profiles | 18 months
  The investigators will compare over time the increase in insulinemia in patients presenting or not the immune activation profile of interest.
Test whether PBMC from patients with Profile#2 induce insulin resistance | 18 months
  The investigators will analyze whether PBMC from patients with the immune activation profile of interest release factors able to inhibit insulin signaling in hepatocytes. Insulin signaling will be measured by quantifying Akt phosphorylation vie western blot.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Eloi Hospital, University Hospital of Montpellier, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Psomas C, Younas M, Reynes C, Cezar R, Portales P, Tuaillon E, Guigues A, Merle C, Atoui N, Fernandez C, Le Moing V, Barbuat C, Marin G, Nagot N, Sotto A, Eliaou JF, Sabatier R, Reynes J, Corbeau P. One of the immune activation profiles observed in HIV-1-infected adults with suppressed viremia is linked to metabolic syndrome: The ACTIVIH study. EBioMedicine. 2016 Jun;8:265-276. doi: 10.1016/j.ebiom.2016.05.008. Epub 2016 May 10. PMID 27428436
- [Derived] Younas M, Gimenez S, Lin YL, Mettling C, Maiorano D, Reynes J, Pasero P, Rondard P, Psomas CK, Corbeau P. gamma-Aminobutyric Acid-Induced Monocytic Reactive Oxygen Species Impair CD4 Restoration in Treated Adults With HIV-1. J Infect Dis. 2025 Jun 2;231(5):1246-1257. doi: 10.1093/infdis/jiaf058. PMID 39903648